CLINICAL TRIAL: NCT01923155
Title: Safety & Effectiveness of Nurse Performed Colonoscopies Under Supervision: A Randomized Controlled Study in Asia (NE Study)
Brief Title: Safety & Effectiveness of Nurse Performed Colonoscopies Under Supervision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Aric Josun Hui, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NE
Record Dates: First submitted 2013-08-12; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Nurse endoscopists (Active Comparator): Colonoscopy performed by nurse endoscopists supervised by senior medical endoscopists
  Interventions: Procedure: Colonoscopy
- Medical endoscopists (Active Comparator): Colonoscopy performed by senior medical endoscopists
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy

SUMMARY:
There is no theoretical or practical reason why non-medical personnel such as nurses could not be trained to perform diagnostic colonoscopy with comparable proficiency as medical endoscopists. Nurse endoscopists have been widely accepted in the United Kingdom for the past 15 years as a valuable resource to cope with the increasing demand for endoscopic service, in particular diagnostic colonoscopy for colorectal screening. A pilot study performed in Hong Kong in 2008 has shown that endoscopy nurses can be trained to perform diagnostic endoscopy safely and reliably. This study aims to demonstrate that properly trained nurse endoscopists have a comparable proficiency in performing colonoscopy procedures as their medical counterparts.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects receiving screening colonoscopy
* 2. Age ≥ 18
* 3. Informed consent

Exclusion Criteria:

* 1. Subjects have undergone colonoscopy in the past 5 years
* 2. Patients with prior colorectal surgery
* 3. Subjects with a personal history of inflammatory bowel disease, colon adenoma or cancer or family history of Familial Adenomatous Polyposis or Familial non-polyposis syndrome
* 4. Pregnant or lactating women
* 5. Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | Up to 3 months

SECONDARY OUTCOMES:
Cecal intubation RATE | Up to 3 months
Withdrawal time | Up to 3 months
Complication rate | Up to 3 months
Patients pain score | Up to 3 months
Patients overall satisfactory score | Up to 3 months
Cecal intubation TIME | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Endoscopy Unit, Alice Ho Miu Ling Nethersole Hospital, Tai Po, Hong Kong

REFERENCES:
- [Derived] Hui AJ, Lau JY, Lam PP, Chui AO, Fan AS, Lam TY, Tse YK, Tang RS, Ng SC, Wu JC, Ching JY, Wong MC, Chan FK, Sung J. Comparison of colonoscopic performance between medical and nurse endoscopists: a non-inferiority randomised controlled study in Asia. Gut. 2015 Jul;64(7):1058-62. doi: 10.1136/gutjnl-2013-306293. Epub 2014 Dec 18. PMID 25524261